CLINICAL TRIAL: NCT04451551
Title: Myocardial Perfusion Imaging by 15O-H2O PET/CT: Reference Values and Prognostic Value
Brief Title: Myocardial Perfusion Imaging by 15O-H2O PET/CT
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 15O-H2O PET Cohort
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Heart Disease
Keywords: Myocardial Perfusion Imaging; Positron-Emission Tomography; Coronary Artery Disease; Coronary Flow Reserve; Myocardial Blood Flow; Prognosis; Reference Value
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trial will include 5000 patients with evident or suspected ischemic heart disease refered to Department of Nuclear Medicine & PET Centre, Aarhus University Hospital, for perfusion imaging by 15O-H2O PET/CT scan of the heart during rest and stress. The patients will undergo the clinical scan as normal.

Data from the scans will be used to determine reference values of the examination.

Follow up will be done for up to 10 years in regards to major cardiovascular events in order to determine the prognostic value of the scan.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected ischemic heart disease referred for a clinical H2O-PET at Department of Nuclear Medicine and PET Centre, Aarhus University Hospital

Exclusion Criteria:

* Claustrophobia, severe asthma, younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with known or suspected ischemic heart disease referred for a clinical H2O-PET at Department of Nuclear Medicine and PET Centre, Aarhus University Hospital, not meeting any exclusion criteria will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Prognostic value within 10 years | 10 years
  Number of participants who experience a major adverse cardiac event within 10 years of follow-up.

SECONDARY OUTCOMES:
Myocardial blood flow | 5 Years
  The myocardial blood flow of participants assessed by 15O-H2O PET/CT
Coronary flow reserve | 5 Years
  The coronary flow reserve of participants assessed by 15O-H2O PET/CT
Pulmonary transit time | 5 Years
  The pulmonary transit time of participants assessed by 15O-H2O PET/CT
Left ventricular end-systolic volume | 5 Years
  The left ventricular end-systolic volume of participants assessed by 15O-H2O PET/CT
Left ventricular end-diastolic volume | 5 Years
  The left ventricular end-diastolic volume of participants assessed by 15O-H2O PET/CT
Right ventricular end-systolic volume | 5 Years
  The right ventricular end-systolic volume of participants assessed by 15O-H2O PET/CT
Right ventricular end-diastolic volume | 5 Years
  The right ventricular end-diastolic volume of participants assessed by 15O-H2O PET/CT
Immediate coronary angiography followup | 5 years
  Number of participants who undergo coronary angiography within 3 months after primary 15O-H2O PET/CT
Immediate percutaneous coronary intervention (PCI) followup | 5 years
  Number of participants who undergo percutaneous coronary intervention within 3 months after primary 15O-H2O PET/CT
Immediate coronary artery bypass graft (CABG) followup | 5 years
  Number of participants who undergo coronary artery bypass graft within 3 months after primary 15O-H2O PET/CT
Prognostic value within 5 years | 5 years
  Number of participants who experience a major adverse cardiac event within 5 years of follow-up.
Prognostic value within 2 years | 2 years
  Number of participants who experience a major adverse cardiac event within 2 years of follow-up.
Prognostic value within 1 years | 1 years
  Number of participants who experience a major adverse cardiac event within 1 years of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus N, Denmark